CLINICAL TRIAL: NCT02901197
Title: Capnography At the Bedside: Leading Educational Efforts (CapABLE Trial)
Brief Title: Capnography At the Bedside: Leading Educational Efforts
Acronym: CapABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1503015415
Record Dates: First submitted 2016-09-09; First posted 2016-09-15 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Emergency
Keywords: capnography
MeSH Terms: conditions — Emergencies | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education and Reminder (Active Comparator): This arm will consist of participants in a location that receive with web based training and exposure to reminder posters in the workplace.
  Interventions: Behavioral: Education and Reminder Posters
- Policy Change (Active Comparator): This arm's participants will not receive an active intervention (education and reminders), however, policy change will take place in this location.
  Interventions: Other: Policy Change

INTERVENTIONS:
Behavioral: Education and Reminder Posters — See arm description
  Arms: Education and Reminder
Other: Policy Change — See arm description
  Arms: Policy Change

SUMMARY:
The purpose of this dual-site quasi-experimental pilot study is to evaluate if the implementation of an educational intervention paired with an environmental assessment to address accessibility barriers is associated with improvement in staff knowledge and skills, and adherence to national guidelines for use (evaluation in the knowledge transfer framework) in an emergency department (ED) setting.

DETAILED DESCRIPTION:
The objective of this study is to develop a multi-faceted implementation program (referred to as the Capnography At the Bedside: Leading Emergency Education (CapABLE Trial)) to increase the use of capnography during two critical events in the emergency department, intubation and CPR, for better detection of endotracheal intubation, endotracheal tube dislodgement, and quality CPR.

The specific aims of the proposed study are to examine:

1. the effect of a comprehensive theory-based educational intervention on staff knowledge and skills related to capnography (outcome measure).
2. the effect of a multi-faceted implementation program on the adherence to national guidelines regarding the use of capnography during critical events in the emergency department (process measure).
3. the sustainability of effects of the implementation program on adherence, knowledge and skills (outcome and process measure).

The design and methods of this study are based on the knowledge transfer framework, which dictates identification of the message, target audience, messenger, process and communication, and evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department (ED) staff
* Staff will include registered nurses, respiratory therapists, technical associates, physicians, physician's assistants and advanced practice nurse practitioners who fulfill the majority of their clinical duties in the ED.

Exclusion Criteria:

* Staff who are assigned to work on other units, but who work in the ED on a casual or per diem status will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Average Monitoring Frequency | Pre intervention 3 months and Post intervention about 6 months
  This outcome will reflect the number of patients the staff applied the monitoring to pre and post intervention.

SECONDARY OUTCOMES:
Knowledge | Pre intervention
  A tool will be developed as part of the study to assess knowledge and how that might change over time (from pre to post)
Knowledge | Post intervention (within 1 month of intervention)
  A tool will be developed as part of the study to assess knowledge and how that might change over time (from pre to post)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Langhan, MD, Principal Investigator — Yale University Dept of Pediatrics, Section of Emergency Medicine

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shah R, Streat DA, Auerbach M, Shabanova V, Langhan ML. Improving Capnography Use for Critically Ill Emergency Patients: An Implementation Study. J Patient Saf. 2022 Jan 1;18(1):e26-e32. doi: 10.1097/PTS.0000000000000683. PMID 32175968